CLINICAL TRIAL: NCT05566951
Title: Efficiency of the Technology-Based Psychosocial Empowerment Program for Home Care of Children With Cancer and Their Parents
Brief Title: Technology-Based Psychosocial Empowerment Program for Home Care of Children With Cancer and Their Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Hazal Ozdemir Koyu, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Technology-Based Program
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Child, Only; Empowerment
Keywords: Cancer; Child; Parents; Home-care; Empowerment
MeSH Terms: conditions — Neoplasms; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the research, it was planned to blind the participant and outcome evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): -The experimental group that applied the technology-based psychosocial program
  Interventions: Other: Psychosocial program
- Control group (Other): Control group receiving standard care
  Interventions: Other: Standart care

INTERVENTIONS:
Other: Psychosocial program — A technology-based model-based psychosocial empowerment program will be implemented for parents and children in the control group.
  Other Names: Technology-based psychosocial program
  Arms: Experimental group
Other: Standart care — Parents and children in the intervention group will be applied standard support approaches to be applied in the center where they receive treatment.
  Arms: Control group

SUMMARY:
This research was planned to evaluate the effectiveness of the technology-based psychosocial empowerment program for home care for children aged 8-18 years with cancer and their parents as a parallel-group randomized controlled study design.The required institutional permission and ethics committee approval was received.The study group of the study consisted of 72 children and parents (intervention group [n=36], control group [n=36]). Data were collected using the descriptive features form, the General Self-Efficacy Scale-Pediatric Cancer Version, the State-Trait Anxiety Inventory for Children, the Pediatric Cancer Coping Scale, the General Self-Efficacy Scale for parents, the Problem Solving Inventory, and the Psychological Resilience Scale for Parents of Children with Cancer. The data were stored in the SPSS 25 program.

DETAILED DESCRIPTION:
The incidence of childhood cancers has become an important health problem increasing all over the world. Children and parents are affected in many dimensions physically, psychologically, and socially during this experience. The needs of the child and parents are not limited to the treatment period in the hospital. They also need to be supported and strengthened during the home care process. The required institutional permission and ethics committee approval was received. The study group of study consisted of 72 children and parents (intervention group [n=36], control group [n=36]).The technology-based program was applied to children and families for 4-6 weeks through modules on the website. In addition, at the end of each module, online interviews or telephone counseling will be applied.Children and parents in the control group will follow the standard care procedures included in the treatment process. At the end of the study, it was planned to apply website modules to the children and parents in the control group. The research is based on the Psychological Empowerment Theory.

ELIGIBILITY:
Inclusion Criteria:

* For children's:
* Children between the ages of 8-18,
* Those receiving cancer treatment (leukemias and solid tumors) and completing the first 2 months of the treatment process,
* Children with tablets, android phones and internet access
* Children whose parents and themselves agree to participate in the study,
* Children who can continue the study for 4-6 weeks,
* For primary care parents,
* Parents who can speak Turkish,
* Parents who can use computers and android mobile phones,
* Parents who agreed to participate in the study,
* Parents who can continue the study for 4-6 weeks,

Exclusion Criteria:

* Newly diagnosed children (in induction phase),
* Children who are in the terminal period or who are treated for relapse,
* Presence of another important disease (such as chronic disease, psychiatric diagnosis) in the family that may prevent coping, other than the child followed up with the diagnosis of cancer

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
General Self-Efficacy Scale-Pediatric Cancer Version | Change from Baseline level 'Self Efficacy' to 2 months (change is being assessed)
  It is a one-dimensional, 10-item scale used to evaluate self-efficacy in children aged 8-18 years with cancer.As the score obtained from the scale increases, the level of self-efficacy also increases.
State-Trait Anxiety Inventory for Children | Change from Baseline level 'State-Trait Anxiety' to 2 months (change is being assessed)
  he 'State-Trait Anxiety Scale' for children between the ages of 8-18 was created to determine what the child feels at that moment, and the 'Stait-Trait Anxiety Scale' was created to determine what they usually feel. The higher the score, the higher the anxiety level.
Pediatric Cancer Coping Scale | Change from Baseline level 'Pediatric Cancer Coping Scale' to 2 months (change is being assessed)
  It was developed to evaluate coping in children aged 7-18 years with cancer diagnosis. The scale consists of 3 sub-dimensions as cognitive coping, problem-focused coping and defensive coping. The higher the score, the higher the coping strategies.
General Self-Efficacy Scale | Change from Baseline level 'Self Efficacy' to 2 months (change is being assessed)
  It is a one-dimensional scale developed to evaluate the general self-efficacy level of adults.As the score obtained from the scale increases, the level of self-efficacy also increases.
Problem Solving Inventory | Change from Baseline level 'Problem Solving Inventory' to 2 months (change is being assessed)
  It is a scale that measures the problem solving skills of individuals according to the perception of the individual.The inventory consists of three sub-dimensions: Safe in Problem Solving, Approach Avoidance Style and Personal Control.Low scores from the inventory indicate the ability to produce effective solutions to problems, while high scores indicate the inability to find effective solutions to problems.
Psychological Resilience Scale for Parents of Children with Cancer | Change from Baseline level 'Psychological Resilience Scale for Parents of Children with Cancer'' to 2 months (change is being assessed)
  The Resilience Scale for Parents of Children was developed to examine the resilience status of parents of children aged 0-18 years with cancer diagnosis. The scale consists of 24 items and 4 sub-dimensions. As the score obtained from the scale increases, the level of psychological resilience of the parents increases.

SECONDARY OUTCOMES:
SSPedi: Symptom Screening Scale in Pediatric Patients | While the intervention continues (1 months), the log records of the scale on the website will be evaluated.
  The screening tool includes 15 symptoms that evaluate the symptoms children have experienced in the last two days. Each symptom is evaluated with a 5-point Likert-type scoring system, and the score range varies between 0-60. Higher scores indicate that the number of symptoms and the discomfort they cause increase

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers.